CLINICAL TRIAL: NCT02742688
Title: Effect of Intake of Pyrus Pyrifolia Var. Culta(Makino) NaKai Peel Extract on Body Fat and Blood Lipid.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yongsoon Park, professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GFB-BF-PE
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyrus pyrifolia var. culta(Makino) NaKai peel extract (Experimental)
  Interventions: Dietary Supplement: Pyrus pyrifolia var. culta(Makino) NaKai peel extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pyrus pyrifolia var. culta(Makino) NaKai peel extract — Pyrus pyrifolia var. culta(Makino) NaKai peel extract(4g/day)
  Arms: Pyrus pyrifolia var. culta(Makino) NaKai peel extract
Dietary Supplement: Placebo — Placebo(4g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Pyrus pyrifolia var. culta(Makino) NaKai peel extract on decrement of body fat. The investigators measured decrement of body fat parameters , including Body Fat Mass, Percent Body Fat, weight and BMI(body mass index), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-65 years old
* BMI(body mass index) 25~29.9 kg/m^2 or WC(Waist Circumference) ≥ 90(men), WC ≥ 85(women)
* Able to give informed consent

Exclusion Criteria:

* BMI(body mass index) ≥ 30 kg/m^2
* Significant variation in weight(more 10%) in the past 3 months
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Changes in body fat mass | 8 week
  Body fat mass was measured in study baseline and visit 3(8 week)

SECONDARY OUTCOMES:
Changes in percent body fat | 8 week
  Percent body fat was measured in study baseline and visit 3(8 week)
Change in fat free mass | 8 week
  Fat free mass was measured in study baseline and visit 3(8week)
Change in body mass index | 8 week
  Body mass index was measured in study baseline and visit 3(8 week)
Change in weight | 8 week
  Weight was measured in study baseline and visit 3(8 week)
Change in total cholesterol | 8 week
  Total cholesterol was measured in study baseline and visit 3(8 week)
Change in triglyceride | 8 week
  Triglyceride was measured in study baseline and visit 3(8 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided